CLINICAL TRIAL: NCT01348438
Title: Transapical Implantation of the Medtronic Engager Transcatheter Aortic Valve Implantation System - The Engager European Pivotal Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG CIP-001
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Aortic Valve Stenosis
Keywords: high risk; surgical valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Other)
  Interventions: Device: Medtronic Engager Transcatheter Aortic Valve Implantation System

INTERVENTIONS:
Device: Medtronic Engager Transcatheter Aortic Valve Implantation System — Transapical implantation of the Medtronic Engager Transcatheter Aortic Valve Implantation System

SUMMARY:
The purpose of the study is to evaluate the safety and clinical performance of the Engager Transcatheter Aortic Valve Implantation System in patients with severe aortic valve stenosis who are at high risk for surgical valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis defined as one or more of the following by Doppler echocardiography: mean gradient > 40 mmHg; max velocity > 4m/s; aortic valve area ≤ 0.8 cm2.
2. Symptoms related to aortic valve disease, and NYHA Functional Class II or greater.
3. Logistic EuroSCORE predicted risk for mortality of ≥20%, or comorbidity judged by the investigator to pose an absolute or relative contraindication for conventional aortic valve replacement.
4. Patient is indicated for aortic valve implantation with a biological prosthesis (tissue valve) in accordance with the 2007 European Society of Cardiology (ESC) Guidelines for management of valvular heart disease.
5. Age ≥ 18 years.
6. Echocardiographically determined aortic annulus diameter of ≥19 mm and ≤ 26 mm in a long-axis view.

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve.
2. Severe eccentricity of calcification, defined as calcium deposits larger than 6mm in diameter.
3. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
4. Left ventricular ejection fraction < 25%, as determined by contrast ventriculography, or echocardiography or radionuclide angiography if contrast ventriculography not available
5. Hypertrophic obstructive cardiomyopathy.
6. Patients with life expectancy less than 12 months due to an underlying non-cardiac comorbid disease.
7. Known hypersensitivity or contraindication that cannot be adequately controlled with pre-medication to any study medication or material, such as contrast medium or Nitinol.
8. Sepsis or acute endocarditis.
9. Blood dyscrasia such as acute anemia, leucopenia, or thrombocytopenia; bleeding diathesis, or coagulopathy.
10. Renal insufficiency assessed by creatinine > 2.5 mg/dl and/or end stage renal disease requiring chronic dialysis.
11. Active peptic ulcer or GI bleeding within 3 months from the planned index procedure.
12. Untreated clinically significant coronary artery disease requiring revascularization.
13. Cardiogenic shock, suspected cardiogenic shock, or hemodynamic instability requiring inotropic support or mechanical heart assistance.
14. Significant aortic disease, including abdominal and thoracic aortic aneurysm, defined as maximal luminal diameter of 5 cm or greater.
15. Need for emergency surgery, cardiac or non-cardiac.
16. History of myocardial infarction in the last 6 weeks.
17. History of TIA or CVA in the last 6 months.
18. Therapeutic invasive cardiac procedure, with the exception of aortic balloon valvuloplasty, performed within 30 days of the planned date of valve implantation, or 6 months in the case of drug-eluting stents.
19. Pre-existing prosthetic heart valve or prosthetic ring in any position.
20. Mitral regurgitation greater than 2+ by angiography or moderate by echocardiography.
21. Patient refuses a blood transfusion.
22. Patient is currently enrolled in another investigational device or drug trial that may influence the outcome of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 Days
  All-cause mortality within 30 days post-implantation

SECONDARY OUTCOMES:
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) free survival at 30 days and 6 months post implantation | 6 months
Device and procedure related Major Adverse Events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Volkmar Falk, Prof., Principal Investigator — University of Zurich; Jean-Louis Vanoverschelde, Prof., Principal Investigator — Cliniques Universitaires Saint-Luc, Brussels
Locations (9):
- Cliniques Universitaires Saint- Luc, Brussels, Belgium
- Germany (6):
  - Kerckhoff-Klinik, Bad Nauheim
  - Ruhr-Universität Bochum, Bad Oeynhausen
  - Uniklinik Köln Heart Center, Cologne
  - Universitätsklinikum Hamburg- Eppendorf, Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München, München
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel
- University of Zurich - Klinik für Herzchirurgie, UniversitätsSpital, Zurich, Switzerland

REFERENCES:
- [Derived] Holzhey D, Linke A, Treede H, Baldus S, Bleiziffer S, Wagner A, Borgermann J, Scholtz W, Vanoverschelde JL, Falk V. Intermediate follow-up results from the multicenter engager European pivotal trial. Ann Thorac Surg. 2013 Dec;96(6):2095-100. doi: 10.1016/j.athoracsur.2013.06.089. Epub 2013 Sep 7. PMID 24021766